CLINICAL TRIAL: NCT00388596
Title: An Open-Label, Partially Randomized, Interaction Study to Evaluate the Effects of SB-751689 on the Pharmacokinetics of Rosuvastatin and Atorvastatin or the Effects of Ketoconazole on the Pharmacokinetics of SB-751689 in Healthy Postmenopausal Female Subjects
Brief Title: A Study Of SB-751689, Atorvastatin, Ketoconazole, And Rosuvastatin In Health Postmenopausal Women.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR9108985
Record Dates: First submitted 2006-10-13; First posted 2006-10-17 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Osteoporosis
Keywords: SB-751689; osteoporosis; drug interaction; ketoconazole; atorvastatin; rosuvastatin
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: SB-751689

SUMMARY:
The first purpose of this study is to determine if taking SB-751689 along with Rosuvastatin (CRESTOR) or Atorvastatin (LIPITOR) will change how Rosuvastatin or Atorvastatin are absorbed and eliminated from the body. Rosuvastatin and Atorvastatin are prescription medications used to treat patients with high cholesterol. Patients who would take SB-751689 for osteoporosis might also take Rosuvastatin or Atorvastatin for high cholesterol. In an earlier study, SB-751689 was shown to lower the blood levels of Rosuvastatin when the two drugs were taken at the same time. Lower blood levels of Rosuvastatin could mean that it would not be as effective in lowering cholesterol. In this study SB-751689 will be taken alone, Rosuvastatin will be taken alone, SB-751689 and Rosuvastatin will be taken together, and SB-751689 will be taken 12 hours before Rosuvastatin is taken. This study will help determine if the two drugs should be taken 12 hour apart to prevent lower Rosuvastatin blood levels. Atorvastatin will be taken alone and at the same time as SB-751689 to determine if Atorvastatin blood levels are lower when taken at the same time as SB-751689.

A second purpose of this study is to determine if taking another drug called Ketoconazole (Nizoral) along with SB-751689 will change how SB-751689 is absorbed and eliminated from the body. Ketoconazole is a prescription medication used to treat patients with fungal and yeast infections.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ambulatory postmenopausal woman defined as being amenorrheic for at least 2 years
* Non-smoker
* Weight >110 lbs (>50 kg)
* Body mass index within the range 19 - 29.9 kg/m2
* are capable of giving written informed consent

Exclusion Criteria:

* Have any clinically relevant abnormality identified on the screening history and physical or laboratory examination, 12-lead surface electrocardiogram (ECG) and/or 24 hour Holter, including QTc > 450 msec
* Test positive urine drug screen or alcohol
* Test positive for HIV, hepatitis B virus or hepatitis C virus
* Smoker or have a history of smoking or use of nicotine containing products within one year of the study or >10 pack-year history of smoking overall
* have a history of regular alcohol consumption exceeding 7 units/week (1 unit = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening
* have a history of drug abuse within 6 months of the study
* have participated in a trial with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication
* use of prescription or non-prescription drugs (including calcium tablets, calcium containing antacids, aspirin or nonsteroidal anti-inflammatory drugs), vitamins, herbal and dietary supplements, within 14 days prior to the first dose of study medication.
* have consumed of grapefruit containing products within 14 days prior to the first dose of study medication
* have donated of blood in excess of 500 mL within 56 days prior to dosing
* have evidence of kidney or liver disease
* have a history of significant gastrointestinal disease or a gastrointestinal surgical procedures
* are sensitive to any of the study medications or components thereof
* have a history of cardiovascular disease
* have medical conditions which might alter bone metabolism
* have a serum parathyroid hormone (iPTH) test, or vitamin D levels outside the normal range

Max Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-10

PRIMARY OUTCOMES:
AUC and Cmax of SB-751689, rosuvastatin, and atorvastatin in blood or plasma. | throughout the study

SECONDARY OUTCOMES:
AUC and Cmax of 2 metabolites of atorvastatin and PTH in plasma. | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MBChB, FRCP, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Miami, Florida, United States